CLINICAL TRIAL: NCT00638014
Title: A Randomized, Controlled, Phase 4 Study of Sternal Plating (Rapid Sternal Closure System, KLS Martin L.P.) in Cardiac Surgical Subjects at Higher Risk for Sternal Wound Complications.
Brief Title: Rapid Sternal Closure System (TALON)
Acronym: TALON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: KLS Martin, L.P. (Unknown)
Responsible Party: Gary Moore/ Regulatory Affair, Quality Assurance, KLS Martin, L.P.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00006260
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Sternal Wound Infection; Mediastinitis
Keywords: Sternal wound closure; cardiac surgery; sternal nonunion
MeSH Terms: conditions — Mediastinitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Conventional wires only
  Interventions: Device: Conventional wire closure
- 2 (Experimental): Rapid Sternal Closure System supplemented with wires
  Interventions: Device: Rapid Sternal Closure System

INTERVENTIONS:
Device: Rapid Sternal Closure System — Sternal talons will be used and supplemented with wires
  Arms: 2
Device: Conventional wire closure — Conventional wire closure of sternum
  Arms: 1

SUMMARY:
The primary objective is to establish if the Rapid Sternal Closure System (RSCS) improves early postoperative recovery as manifested by decreased pain and improved pulmonary function.

Secondary objectives include evaluation of Rapid Sternal Closure System with regard to SWCs (surgical wound complication defined as surgically treated sternal wound infection and sternal instability/non-union) as outlined in the protocol.

For a given study endpoint, the null hypothesis will be no difference between the Rapid Sternal Closure System group and the control group. The alternative hypothesis will be a difference between 2 groups. The statistical objective of this study is to reject the null hypothesis in favor of the alternative hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. Women of childbearing potential must have a negative serum (or urine) human chorionic gonadotropin assay prior to surgery, and be willing to continue to use effective means of birth control for at least 180 days following surgery. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B(TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use.
2. Age ≥ 18 years.
3. Scheduled to undergo nonemergent on or off pump coronary artery bypass graft (CABG) and/or valve repair or replacement surgery through a full median sternotomy.
4. At higher risk for SWC, defined as the presence of any of the following factors: obesity (body mass index > 30), chronic steroid use (>6 month duration and currently using), severe chronic obstructive pulomonary disease, planned bilateral internal mammary artery harvest, undergoing redo median sternotomy, and history of radiation to the chest.
5. Willing and able to provide written informed consent.
6. Available for evaluation from baseline until final evaluation at 180 days postsurgery.

Exclusion Criteria:

1. Undergoing emergency cardiac surgery (urgent surgery is allowed if informed consent is obtained and the study procedures can be performed).
2. Undergoing a significant concomitant surgical procedure (eg, carotid endarterectomy, aortic root repair or replacement, deep hypothermic circulatory arrest [DHCA], or pulmonary resection).
3. Undergoing a minimally invasive or a thoracic surgical approach.
4. Using a preoperative mechanical assist device or intraaortic balloon pump (IABP), if inserted for shock/low output syndrome (an IABP is allowed if it is inserted for unstable angina or low ejection fraction).
5. Active and significant systemic infection, eg, active endocarditis or a history of significant recurrent systemic infection.
6. Receiving antibiotic therapy within the 2 weeks before the date of surgery.
7. History of malignancy within the past year (except for squamous or basal cell carcinoma of the skin that has been treated, with no evidence of recurrence).
8. History of major organ transplantation, including bone marrow transplantation.
9. Recent history of significant drug or alcohol abuse.
10. Current immunosuppressive condition (eg, symptomatic human immunodeficiency virus [HIV] infection). Use of steroids is not an exclusion criteria).
11. Female subject who is pregnant (including a positive pregnancy test at screening or baseline) or nursing. Females of childbearing potential not practicing a birth control method with a high degree of reliability.
12. Postsurgical life expectancy ≤ 90 days, in the investigator's or sponsor's opinion.
13. Current participation or participation within 30 days before the start of this study in an experimental drug or device study or currently participating in a study during which the administration of investigational drugs within 90 days is anticipated.
14. Refusal to accept medically indicated blood products.
15. Moderate or severe pectus deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Bennett-Guerrero, M. D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Fry DE. The economic costs of surgical site infection. Surg Infect (Larchmt). 2002;3 Suppl 1:S37-43. doi: 10.1089/sur.2002.3.s1-37. PMID 12573038
- [Background] Friberg O, Dahlin LG, Levin LA, Magnusson A, Granfeldt H, Kallman J, Svedjeholm R. Cost effectiveness of local collagen-gentamicin as prophylaxis for sternal wound infections in different risk groups. Scand Cardiovasc J. 2006 Apr;40(2):117-25. doi: 10.1080/14017430500363024. PMID 16608782
- [Background] Demmy TL, Park SB, Liebler GA, Burkholder JA, Maher TD, Benckart DH, Magovern GJ Jr, Magovern GJ Sr. Recent experience with major sternal wound complications. Ann Thorac Surg. 1990 Mar;49(3):458-62. doi: 10.1016/0003-4975(90)90256-6. PMID 2310254
- [Background] Tang GH, Maganti M, Weisel RD, Borger MA. Prevention and management of deep sternal wound infection. Semin Thorac Cardiovasc Surg. 2004 Spring;16(1):62-9. doi: 10.1053/j.semtcvs.2004.01.005. PMID 15366689
- [Background] Braxton JH, Marrin CA, McGrath PD, Morton JR, Norotsky M, Charlesworth DC, Lahey SJ, Clough R, Ross CS, Olmstead EM, O'Connor GT. 10-year follow-up of patients with and without mediastinitis. Semin Thorac Cardiovasc Surg. 2004 Spring;16(1):70-6. doi: 10.1053/j.semtcvs.2004.01.006. PMID 15366690
- [Background] Hollenbeak CS, Murphy DM, Koenig S, Woodward RS, Dunagan WC, Fraser VJ. The clinical and economic impact of deep chest surgical site infections following coronary artery bypass graft surgery. Chest. 2000 Aug;118(2):397-402. doi: 10.1378/chest.118.2.397. PMID 10936131
- [Background] Boyce JM, Potter-Bynoe G, Dziobek L. Hospital reimbursement patterns among patients with surgical wound infections following open heart surgery. Infect Control Hosp Epidemiol. 1990 Feb;11(2):89-93. doi: 10.1086/646127. PMID 2107250
- [Background] Baskett RJ, MacDougall CE, Ross DB. Is mediastinitis a preventable complication? A 10-year review. Ann Thorac Surg. 1999 Feb;67(2):462-5. doi: 10.1016/s0003-4975(98)01195-3. PMID 10197671
- [Background] Sakamoto H, Fukuda I, Oosaka M, Nakata H. Risk factors and treatment of deep sternal wound infection after cardiac operation. Ann Thorac Cardiovasc Surg. 2003 Aug;9(4):226-32. PMID 13129420
- [Background] Crabtree TD, Codd JE, Fraser VJ, Bailey MS, Olsen MA, Damiano RJ Jr. Multivariate analysis of risk factors for deep and superficial sternal infection after coronary artery bypass grafting at a tertiary care medical center. Semin Thorac Cardiovasc Surg. 2004 Spring;16(1):53-61. doi: 10.1053/j.semtcvs.2004.01.009. PMID 15366688
- [Background] Fowler VG Jr, O'Brien SM, Muhlbaier LH, Corey GR, Ferguson TB, Peterson ED. Clinical predictors of major infections after cardiac surgery. Circulation. 2005 Aug 30;112(9 Suppl):I358-65. doi: 10.1161/CIRCULATIONAHA.104.525790. PMID 16159846
- [Background] Olsen MA, Lock-Buckley P, Hopkins D, Polish LB, Sundt TM, Fraser VJ. The risk factors for deep and superficial chest surgical-site infections after coronary artery bypass graft surgery are different. J Thorac Cardiovasc Surg. 2002 Jul;124(1):136-45. doi: 10.1067/mtc.2002.122306. PMID 12091819
- [Background] Ridderstolpe L, Gill H, Granfeldt H, Ahlfeldt H, Rutberg H. Superficial and deep sternal wound complications: incidence, risk factors and mortality. Eur J Cardiothorac Surg. 2001 Dec;20(6):1168-75. doi: 10.1016/s1010-7940(01)00991-5. PMID 11717023
- [Background] Trick WE, Scheckler WE, Tokars JI, Jones KC, Reppen ML, Smith EM, Jarvis WR. Modifiable risk factors associated with deep sternal site infection after coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2000 Jan;119(1):108-14. doi: 10.1016/s0022-5223(00)70224-8. PMID 10612768
- [Background] Abboud CS, Wey SB, Baltar VT. Risk factors for mediastinitis after cardiac surgery. Ann Thorac Surg. 2004 Feb;77(2):676-83. doi: 10.1016/S0003-4975(03)01523-6. PMID 14759458
- [Background] Dodds Ashley ES, Carroll DN, Engemann JJ, Harris AD, Fowler VG Jr, Sexton DJ, Kaye KS. Risk factors for postoperative mediastinitis due to methicillin-resistant Staphylococcus aureus. Clin Infect Dis. 2004 Jun 1;38(11):1555-60. doi: 10.1086/420819. Epub 2004 May 12. PMID 15156442
- [Background] Lu JC, Grayson AD, Jha P, Srinivasan AK, Fabri BM. Risk factors for sternal wound infection and mid-term survival following coronary artery bypass surgery. Eur J Cardiothorac Surg. 2003 Jun;23(6):943-9. doi: 10.1016/s1010-7940(03)00137-4. PMID 12829070
- [Background] Jonkers D, Elenbaas T, Terporten P, Nieman F, Stobberingh E. Prevalence of 90-days postoperative wound infections after cardiac surgery. Eur J Cardiothorac Surg. 2003 Jan;23(1):97-102. doi: 10.1016/s1010-7940(02)00662-0. PMID 12493512
- [Background] Eklund AM, Valtonen M, Werkkala KA. Prophylaxis of sternal wound infections with gentamicin-collagen implant: randomized controlled study in cardiac surgery. J Hosp Infect. 2005 Feb;59(2):108-12. doi: 10.1016/j.jhin.2004.10.005. PMID 15620444
- [Background] Finkelstein R, Rabino G, Mashiah T, Bar-El Y, Adler Z, Kertzman V, Cohen O, Milo S. Vancomycin versus cefazolin prophylaxis for cardiac surgery in the setting of a high prevalence of methicillin-resistant staphylococcal infections. J Thorac Cardiovasc Surg. 2002 Feb;123(2):326-32. doi: 10.1067/mtc.2002.119698. PMID 11828293
- [Background] Friberg O, Svedjeholm R, Soderquist B, Granfeldt H, Vikerfors T, Kallman J. Local gentamicin reduces sternal wound infections after cardiac surgery: a randomized controlled trial. Ann Thorac Surg. 2005 Jan;79(1):153-61; discussion 161-2. doi: 10.1016/j.athoracsur.2004.06.043. PMID 15620935
- [Background] Dickie SR, Dorafshar AH, Song DH. Definitive closure of the infected median sternotomy wound: a treatment algorithm utilizing vacuum-assisted closure followed by rigid plate fixation. Ann Plast Surg. 2006 Jun;56(6):680-5. doi: 10.1097/01.sap.0000202825.41069.c3. PMID 16721085
- [Background] Hendrickson SC, Koger KE, Morea CJ, Aponte RL, Smith PK, Levin LS. Sternal plating for the treatment of sternal nonunion. Ann Thorac Surg. 1996 Aug;62(2):512-8. PMID 8694615
- [Background] Pai S, Gunja NJ, Dupak EL, McMahon NL, Roth TP, Lalikos JF, Dunn RM, Francalancia N, Pins GD, Billiar KL. In vitro comparison of wire and plate fixation for midline sternotomies. Ann Thorac Surg. 2005 Sep;80(3):962-8. doi: 10.1016/j.athoracsur.2005.03.089. PMID 16122464
- [Background] Song DH, Lohman RF, Renucci JD, Jeevanandam V, Raman J. Primary sternal plating in high-risk patients prevents mediastinitis. Eur J Cardiothorac Surg. 2004 Aug;26(2):367-72. doi: 10.1016/j.ejcts.2004.04.038. PMID 15296898
- [Background] Edwards FH, Engelman RM, Houck P, Shahian DM, Bridges CR; Society of Thoracic Surgeons. The Society of Thoracic Surgeons Practice Guideline Series: Antibiotic Prophylaxis in Cardiac Surgery, Part I: Duration. Ann Thorac Surg. 2006 Jan;81(1):397-404. doi: 10.1016/j.athoracsur.2005.06.034. No abstract available. PMID 16368422
- [Background] Bratzler DW, Houck PM; Surgical Infection Prevention Guidelines Writers Workgroup; American Academy of Orthopaedic Surgeons; American Association of Critical Care Nurses; American Association of Nurse Anesthetists; American College of Surgeons; American College of Osteopathic Surgeons; American Geriatrics Society; American Society of Anesthesiologists; American Society of Colon and Rectal Surgeons; American Society of Health-System Pharmacists; American Society of PeriAnesthesia Nurses; Ascension Health; Association of periOperative Registered Nurses; Association for Professionals in Infection Control and Epidemiology; Infectious Diseases Society of America; Medical Letter; Premier; Society for Healthcare Epidemiology of America; Society of Thoracic Surgeons; Surgical Infection Society. Antimicrobial prophylaxis for surgery: an advisory statement from the National Surgical Infection Prevention Project. Clin Infect Dis. 2004 Jun 15;38(12):1706-15. doi: 10.1086/421095. Epub 2004 May 26. PMID 15227616
- [Background] Engelman R, Shahian D, Shemin R, Guy TS, Bratzler D, Edwards F, Jacobs M, Fernando H, Bridges C; Workforce on Evidence-Based Medicine, Society of Thoracic Surgeons. The Society of Thoracic Surgeons practice guideline series: Antibiotic prophylaxis in cardiac surgery, part II: Antibiotic choice. Ann Thorac Surg. 2007 Apr;83(4):1569-76. doi: 10.1016/j.athoracsur.2006.09.046. No abstract available. PMID 17383396
- [Background] Bolon MK, Morlote M, Weber SG, Koplan B, Carmeli Y, Wright SB. Glycopeptides are no more effective than beta-lactam agents for prevention of surgical site infection after cardiac surgery: a meta-analysis. Clin Infect Dis. 2004 May 15;38(10):1357-63. doi: 10.1086/383318. Epub 2004 Apr 21. PMID 15156470
- [Background] Harton SC, Grap MJ, Savage L, Elswick RK. Frequency and predictors of return to incentive spirometry volume baseline after cardiac surgery. Prog Cardiovasc Nurs. 2007 Winter;22(1):7-12. doi: 10.1111/j.0889-7204.2007.05199.x. PMID 17342000
- [Background] Dhadwal K, Al-Ruzzeh S, Athanasiou T, Choudhury M, Tekkis P, Vuddamalay P, Lyster H, Amrani M, George S. Comparison of clinical and economic outcomes of two antibiotic prophylaxis regimens for sternal wound infection in high-risk patients following coronary artery bypass grafting surgery: a prospective randomised double-blind controlled trial. Heart. 2007 Sep;93(9):1126-33. doi: 10.1136/hrt.2006.103002. Epub 2007 Feb 19. PMID 17309908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented and enrolled in the study at 2 centers from April 2008 to July 2009.
Pre-assignment Details: Overall 53 subjects were consented and enrolled in the study from April 2008 to July 2009. Two patients were not included in the analysis (1 patients' surgery was cancelled, 1 patient was not randomized due to logistical reasons), leaving a total of 51 subjects who were included in the modified intent-to-treat analysis.
Groups:
- Conventional Wires Only: The control group received conventional wires including double wires to close the sternum.
- Talon: Subjects randomized to the Talon group received Talons in the sternum plus supplementary wires in the manubrium. The number of Talons inserted was based on patient factors/clinician judgment. For study subjects randomized to the Talon, the device was to be inserted/used in an identical manner to use of the Talon in non-study patients.
Period: Overall Study
Arm/Group | Conventional Wires Only | Talon
Started | 23 | 28
Completed | 23 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Wires Only | Talon | Total
Number analyzed (Participants) | 23 | 28 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 9 | 12 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.2) | 61.8 (10.0) | 62.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 14 | 24 | 38
Region of Enrollment [Number; unit: participants]
  United States | 23 | 28 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of Preoperative Incentive Spirometry (IS) Volume Achieved
Description: Maximum incentive spirometry volume was measured at baseline (prior to surgery) and daily from postoperative day 1 through postoperative day 7 (or discharge if earlier) using a Coach 2 incentive spirometer with one way valve (Coach 2 model # 22-4000, Smiths Medical, Keene, NH).
Time Frame: Baseline, Maximum value during postoperatively days 1 thru 7
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Conventional Wires Only | Talon
Number analyzed (Participants) | 23 | 28
percentage change | 58 (24) | 67 (32)
Statistical Analysis 1: Comparison: Conventional Wires Only vs Talon; Test type: Superiority or Other; p = 0.41, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Sternal Wound Infection or Sternal Instability/Non-union
Description: The Data and Safety Monitoring Board reviewed source documents for all cases with possible sternal wound infection and sternal instability or non-union and made a determination as to the presence of these complications.
Time Frame: Up to 180 days
Measure: Number; unit: Participants
Arm/Group | Conventional Wires Only | Talon
Number analyzed (Participants) | 23 | 28
Participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Conventional Wires Only | Talon
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/28
Other Adverse Events (participants affected / at risk) | 0/23 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Wires Only (N=23) | Talon (N=28)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Randomized to Standard of Care arm
Chest tube entrapment between sternal halves (not Talon) (Surgical and medical procedures) | 0 (0) | 1 (1) — Chest tube entrapped between sternal halves, but not Talon device. Surgeon considered this NOT related to study. DSMB reviewed event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No